CLINICAL TRIAL: NCT07244081
Title: Effects of Kinesiotherapy on Upper Limb Function and Activities of Daily Living in Children With Hemiplegic Cerebral Palsy
Brief Title: Kinesiotherapy on Upper Limb Function and Activities of Daily Living in Children With Hemiplegic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/RCR&AHS/NAIMAANDLEEB
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Kinesiotherapy, Hemiplegic Cerebral Palsy, Upper limb function, ADLs
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: . The study will include 28 patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will be age of 8-13 years old of both sexes, ability to follow simple instructions, able to sit or stand with support to participate in physical therapy sessions( MACS level Ⅰ-Ⅲ) and (GMFCS level Ⅰ-Ⅲ), ability to communicate needs and discomfort (verbally or non-verbally), No concurrent participation in other physical therapy and excluded with Severe visual and hearing impairments, severe cognitive disabilities, History of seizures, Recent (within 6 months) or planned orthopedic surgery, Concurrent use of botulinum toxin injections. Experimental group will perform both Kinesiotherapy protocol and conventional physical therapy while Control group will perform only conventional physical therapy for 8 weeks 2-3 times weekly with 45 min of each session. Outcomes to be analyzed will be upper limb function and Activities of daily living (ADLs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Following baseline assessments, participants will begin their respective 8-week intervention program with 2-3 times per week. The group A will receive base line conventional exercise program with standard physical therapy interventions as follow:
  * Stretching of tight muscles of affected upper limb.
  * Weight bearing of affected upper limb.
  * Manual dexterity exercises like grasp release, pack board activities.
  * Teaching of ADLs.
  * Functional task practice(2)
  Interventions: Other: control
- experimental group (Experimental): Kinesiotherapy tailored exercises focusing on movement and exercise, The movements are as follows:Sitting on a chair, the participant had to lean forward to pick up an object previously placed on the floor.Sitting on a chair, the participant had to rotate the upper body, reaching out and grabbing an object on its side, at the height of his shoulders.Sitting on a chair, the participant had to clasp his hands and flex the shoulders.
  Sitting on a chair in front of a table, the participant had to take objects numbered in ascending order and hand them over to the therapist.
  Sitting on a chair holding a stick, the participant had to place one hand above the other, raising his hands as if holding on to the stick.Sitting on a chair in front of a table, the patient had to find similar playing cards. All cards were face down. Sitting on a stretcher, the participant had to laterally tilt his trunk, putting the weight on the upper limbs. The therapist maintained the elbow extension
  Interventions: Other: experimental

INTERVENTIONS:
Other: control — Following baseline assessments, participants will begin their respective 8-week intervention program with 2-3 times per week. The group A will receive base line conventional exercise program with standard physical therapy interventions as follow:
  * Stretching of tight muscles of affected upper limb.
  * Weight bearing of affected upper limb.
  * Manual dexterity exercises like grasp release, pack board activities.
  * Teaching of ADLs.
  * Functional task practice(2)
  Other Names: baseline
  Arms: control group
Other: experimental — Following baseline assessments, participants will begin their respective 8-week intervention program with 2-3 times per week. The group A will receive base line conventional exercise program with standard physical therapy interventions as follow:
  * Stretching of tight muscles of affected upper limb.
  * Weight bearing of affected upper limb.
  * Manual dexterity exercises like grasp release, pack board activities.
  * Teaching of ADLs.
  * Functional task practice(2)
  Other Names: kinesiotherapy
  Arms: experimental group

SUMMARY:
This study will be randomized controlled trial, data will be collected from BASES special education school sialkot , Allama Iqbal Memorial Hospital, sialkot and Lahore. The study will include 28 patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will be age of 8-13 years old of both sexes, ability to follow simple instructions, able to sit or stand with support to participate in physical therapy sessions( MACS level Ⅰ-Ⅲ) and (GMFCS level Ⅰ-Ⅲ), ability to communicate needs and discomfort (verbally or non-verbally), No concurrent participation in other physical therapy and excluded with Severe visual and hearing impairments, severe cognitive disabilities, History of seizures, Recent (within 6 months) or planned orthopedic surgery, Concurrent use of botulinum toxin injections. Experimental group will perform both Kinesiotherapy protocol and conventional physical therapy while Control group will perform only conventional physical therapy for 8 weeks 2-3 times weekly with 45 min of each session. Outcomes to be analyzed will be upper limb function and Activities of daily living (ADLs). Tools used for data collection will be Action Research Arm (ARA) test, Pediatric Evaluation of Disability Inventory (PEDI). Data will be analyzed through SPSS version 26, 27.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a non progressive neurodevelopmental disorder affecting motor function, resulting from damage to the brain. Hemiplegic CP specifically impacting one side of the body with upper extremity generally more effected than the lower. Twenty percent of children with spastic CP have hemiplegia. Upper limb dysfunction and limited activities of daily living (ADLs) significantly impact quality of life, social participation, and independence. Kinesiotherapy, a movement-based therapy that incorporates movements to improve strength, function and mobility. shows promise effects on stroke patients, but its effectiveness on hemiplegic cerebral palsy requires rigorous investigation. This study aims to investigate the effectiveness of kinesiotherapy in improving upper limb function and ADLs in children with hemiplegic cerebral palsy.

This study will be randomized controlled trial, data will be collected from BASES special education school sialkot , Allama Iqbal Memorial Hospital, sialkot and Lahore. The study will include 28 patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will be age of 8-13 years old of both sexes, ability to follow simple instructions, able to sit or stand with support to participate in physical therapy sessions( MACS level Ⅰ-Ⅲ) and (GMFCS level Ⅰ-Ⅲ), ability to communicate needs and discomfort (verbally or non-verbally), No concurrent participation in other physical therapy and excluded with Severe visual and hearing impairments, severe cognitive disabilities, History of seizures, Recent (within 6 months) or planned orthopedic surgery, Concurrent use of botulinum toxin injections. Experimental group will perform both Kinesiotherapy protocol and conventional physical therapy while Control group will perform only conventional physical therapy for 8 weeks 2-3 times weekly with 45 min of each session. Outcomes to be analyzed will be upper limb function and Activities of daily living (ADLs). Tools used for data collection will be Action Research Arm (ARA) test, Pediatric Evaluation of Disability Inventory (PEDI). Data will be analyzed through SPSS version 26, 27.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-13 years old both sexes
* Ability to follow simple instructions, able to sit or stand with support to participate in physical therapy sessions( MACS level Ⅰ-Ⅲ)(9) and (GMFCS level Ⅰ-Ⅲ)(10)
* Ability to communicate needs and discomfort (verbally or non-verbally)
* No concurrent participation in other physical therapy or rehabilitation programs

Exclusion Criteria:

* Severe visual and hearing impairments that would hinder participation
* Severe cognitive or intellectual disabilities that would impede understanding of instructions
* History of seizures or other neurological conditions that may impact participation
* Recent (within 6 months) or planned orthopedic surgery
* Concurrent use of botulinum toxin injections or oral medications affecting muscle tone(2).

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
action arm research arm test | baseline, 8 weeks
  The Action Research Arm Test (ARAT) is a 19 item observational measures used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery, brain injury and multiple sclerosis populations. Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task maximum score 57 means better performance
pediatric evaluation of disability inventory | baseline, 8 weeks
  The PEDI is a standardized clinical assessment tool designed to measure the functional performance of children with typical development whose chronological age is below 7.5 years old, and the functional performance of children with disabilities whose functional capabilities are below those of a 7.5-year-old child. The PEDI can be used for children with developmental disabilities aged 6 months to 21 years and for individuals without disabilities aged less than 7 years(12) The PEDI is composed of 3 domains: functional skill, caregiver assistance, and modification. Each domain includes 3 sub-domains: self-care, mobility, and social function. The functional skill domain, which was used for measuring ADL performance, consists of 197 specific questions. Each child is assigned either 1 point for being capable of performing the assigned task or 0 points for incomplete performance or being unable to perform the task. The reliability of the functional skill subscale of the PEDI is very high.

CONTACTS AND LOCATIONS:
Overall Officials: Naima Andleeb, MS PT, Principal Investigator — Riphah Internatonal university
Locations (1):
- Maria, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberti EJ, Targa ADS, Pichorim SF, Brawerman A. Ludic Table: a comparative study between playful rehabilitation and kinesiotherapy in restricting upper limb movements in individuals with stroke. Med Biol Eng Comput. 2022 Apr;60(4):1187-1198. doi: 10.1007/s11517-022-02532-0. Epub 2022 Mar 4. PMID 35244860